CLINICAL TRIAL: NCT02771886
Title: Evaluation of a Brief "Surf the Urge" Intervention
Brief Title: Evaluation of a Brief Surf the Urge Intervention
Acronym: SUBMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kimberly N Schubert (Other)
Responsible Party: Sponsor-Investigator, Kimberly N Schubert, Doctoral Practicum Student, University of Nevada, Las Vegas
Organization: University of Nevada, Las Vegas (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUBMI-2015
Record Dates: First submitted 2015-12-17; First posted 2016-05-13 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Substance Use; Deliberate Self-harm; Trichotillomania; Aggression; Stealing; Eating Pathology; Gambling
Keywords: mindfulness; urges; adolescents; risk behaviors; therapy intervention
MeSH Terms: conditions — Substance-Related Disorders; Self-Injurious Behavior; Trichotillomania; Aggression; Gambling; Risk-Taking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2-week intervention group (Active Comparator): The "Surf the Urge" intervention will be provided to the participant during his or her 2nd week in the study. The duration of the study will be 6 weeks.
  Interventions: Behavioral: Surf the Urge
- 4-week intervention group (Active Comparator): The "Surf the Urge" intervention will be provided to the participant during his or her 4th week in the study. The duration of the study will be 6 weeks.
  Interventions: Behavioral: Surf the Urge

INTERVENTIONS:
Behavioral: Surf the Urge — The intervention teaches clients to be aware of and accept their feelings, thoughts, and sensations in a non-judgmental manner. Clients learn to remain present within the moment, become aware of their urges, and focus on accepting thoughts and feelings rather than suppressing or changing them. It utilizes visual imagery to assist clients in utilizing more acceptance skills; the client imagines his urges as waves within the ocean and then imagines surfing the waves.
  Some interventionists also provide psychoeducation. Clients learn that urges will not last forever; clients are also taught information about reinforcing urges. The interventionist explains that if clients do not reinforce urges (e.g., do not smoke when an urge to smoke arises) they will eventual subside; however, reinforcing urges (smoke when an urge to smoke arises) will produce stronger urges. Emphasis is placed on the belief that clients have the choice to refrain from engaging in urge-related behaviors.
  Other Names: Surfing the Urge

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a brief "Surf the Urge" intervention to reduce adolescent and young adult (i.e., 14 to 24 years old) urge-related behaviors. These behaviors will include, but not be limited to, substance use, deliberate self-harm, aggressive behavior, pulling out hair, and loosing control when eating.The intervention will utilize mindfulness skills (i.e., awareness, acceptance, nonjudgment) to assist in reducing these risky behaviors.

DETAILED DESCRIPTION:
Empirical research has not specifically examined the effectiveness of the Surf the Urge intervention with an adolescent and young adult sample. Additionally, the value of this intervention with urge-related behaviors besides smoking (e.g., substance use, purging,, deliberate self-harm) is unclear. The current study will examine the efficacy of the Surf the Urge intervention in a sample of 14 to 24-year-olds who engage in a diverse array of urge-related behaviors. To aid participants in reducing their urge-related behavior, and coping with urges, the investigators will cue urges during the intervention by utilizing a cue exposure script. Urge-related behaviors to examine include alcohol use, drug use, tobacco use, deliberate self-harm, and self-induced vomiting. Additionally, only participants who experience urges or engage in the urge-related behavior a minimum of one time per week will be included. If participants report engaging in several urge-related behaviors, or experiencing varying urges, throughout a one-week period, they will be prompted to report the urge engaged in, or experienced, more frequently.purging, restrictive eating, violent actions (e.g., punching someone), gambling, stealing, trichotillomania, etc.

Additionally, the duration of the study will consist of a 6-week time-period, with the intervention occurring at either 2- or 4-weeks, creating a mixed-design model. This model will require fewer participants and allow the evaluation of individual differences related to intervention effectiveness. Additionally, this will enable the comparison of whether participants who were provided with the intervention at 2-weeks, compared to 4-weeks, were able to reduce their urge-related behaviors earlier. It is hypothesized that:

1. The Surf the Urge mindfulness intervention will decrease various urge-related behaviors (e.g., substance use, deliberate self-harm); however, this intervention will not directly affect a participant's self reported urge levels. Furthermore, individuals in the 2- week intervention group will reduce their urge-related behaviors sooner than those in the 4-week intervention group.
2. Participants who score higher on a self-report mindfulness questionnaire (Five Facet Mindfulness Questionnaire) will show greater reductions in their urge-related behaviors (e.g., substance use, deliberate self-harm).
3. Participants who demonstrate the greatest change from their pre- to post- assessment mindfulness self-report scores (Five Facet Mindfulness Questionnaire) will show the greatest changes in urge-related behaviors. They will also rate the Surf the Urge intervention as more satisfying (Client Satisfaction Questionnaire-8).
4. Participants who rate the Surf the Urge intervention as more satisfying (Client Satisfaction Questionnaire-8) will demonstrate a greater reduction in their urge-related behaviors.
5. There will be a 95% adherence rate to both the cue exposure and Surf the Urge protocols demonstrating proper implementation. When assessing intervention integrity, there will be no statistically significant difference in adherence between trained therapists and myself.

This study will provide information on the effectiveness of a brief mindfulness intervention to reduce various urge-related behaviors in a high-risk population (i.e., adolescents). It will provide additional information on a growingly popular intervention technique in a newly studied population and with newly examined problem behaviors. These results may lead to further information on the effectiveness of mindfulness interventions with adolescents and have implications for future treatment modalities. Additionally, it will also provide information on the characteristics of individuals who may be more responsive to briefer urge-behavior reduction interventions.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 14 and 24 years old
* Endorses engaging in an urge-related behavior, or experiencing urges for an urge-related behavior, within the past week
* Currently receiving treatment (or seeking services) at a university mental health clinic at University of Nevada, Las Vegas OR enrolled in a course requiring research participation at University of Nevada, Las Vegas

Exclusion Criteria:

* Younger than 14
* Older than 24
* Does not endorse experiencing urge, or conducting urge-related behavior engagement, during the past week

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change of mindfulness skills from baseline at 6 weeks | week 1 of study duration; week 6 of study duration
  Five Facet Mindfulness Questionnaire. This self-report analysis of trait mindfulness consists of 39 items based on a 5-point Likert scales, ranging from 1 (Never or Very Rarely True) to 5 (Very Often or Always True). Questions assess five factors of mindfulness, including observing, describing, acting with awareness, non-judging of inner experiences, and non-reactivity to inner experiences.
Change of urge feelings from baseline at 6 weeks | each week of the study's duration or once a week for 6 weeks
  The Urge for Urge-Related Behavior Questionnaire (UURBQ) will assess urges for urge-related behavior. Modifying two widely used valid and reliable measures will create this measure. These measures include the extensively utilized Alcohol Urge Questionnaire (AUQ) and Cocaine Craving Questionnaire (CCQ).The UURBQ will leave "a drink" and "cocaine/coke" blank. This will allow me to fill in the blank with the necessary urge-related behavior (e.g., alcohol, illicit substance, cutting) for each participant assessed. There will be 8 items included within this measure. A slight modification of this measure's response scale will occur. Rather than a check mark along a line with a 0 (Strongly Agree) to 100 (Strongly Disagree) based on the AUQ and CCQ, responses will be based on a 7-point Likert Scales ranging from 0 (Strongly Agree) to 7 (Strongly Disagree). This measure will assess urges for numerous urge-related behaviors.
Change in urge-related behavior engagement from baseline at 6 weeks | each week of the study's duration or once a week for 6 weeks
  The Urge-Related Behavior Engagement Questionnaire measure was developed by modifying similar approaches utilized in previous research assessing whether mindfulness interventions reduced an urge-related behavior (e.g., smoking cessation). Participants will report, "How many times have you engaged in [urge-related behavior] during the past week?" I will fill in the blank (i.e., [urge-related behavior]) with the participant's unique urge-related behavior (e.g., alcohol use, illicit drug use, deliberate self-harm) disclosed during the consent procedure. This will ensure that each participant is asked the same question about his or her unique urge-related behavior. Responses will be based on a 6-point Likert scale. The response options will include, 0) not at all, 1) one to two times, 2) three to four times, 3) once per day for all 7 days, 4) more than once per day, but not for all 7 days, 5) more than once per day, on all 7 days.
Client Satisfaction Questionnaire-8 | week 6 of study duration
  This measure consists of 8 items based on a 4-point Likert scales. Each item has a different range 4-point Likert scale response. For example, ranging from 1 (Poor) to 4 (Excellent) or 1(No, Definitely) to 4 (Yes, Definitely).

SECONDARY OUTCOMES:
Demographics | week 1 of study duration
  age, gender, ethnicity, receiving intervention services elsewhere, relationship status
The Multidimensional Personality Questionnaire-Brief Form | week 1 of study duration
  Self-report measure of personality consists of 155, True-False, items. This measure assesses 11 primary subscales of personality, with 12 items each, an Unlikely Virtues subscale that is 14 items, and 9 additional validity items (i.e., VRIN, TRIN). The subscales include: Wellbeing, Social Potency, Achievement, Social Closeness, Stress Reaction, Alienation, Aggression, Control, Harm Avoidance, Traditionalism, and Absorption.
Change in mental health symptoms from baseline at 6 weeks | each week of study's duration or once a week for 6 weeks
  The Depression, Anxiety, and Stress Scale consists of 21 items based on a 4-point Likert scales, ranging from zero (Never or Did Not Apply to Me at All) to 3 (Almost Always or Applied to Me Very Much, or Most of the Time). This measure assesses wellbeing based on the three primary domains of a person's life: depression, anxiety, and stress; consequently, breaking this assessment into three subscales. Each subscale measures various domains of that construct; for example, the depression scale includes an assessment of dysphoria, hopelessness, and anhedonia.

OTHER OUTCOMES:
North American Reading Test | week 1 of study duration
  This measure is comprised of a list of 50 words that increase in difficulty as the assessment progresses. The participant is required to read aloud the list and the researcher records the number of errors made. This assessment evaluates the individual's intelligence (i.e., crystallized intelligence) based on his ability to correctly read and pronounce these 50 words.
Change in risk taking perceptions from baseline at 6 weeks | week 1 of study duration; week 6 of study duration
  This Domain Specific Risk Taking Scale consists of 30 items based on three 7-point Likert scales. The first scale asks participants how likely they are to engage in the behavior ranging from 1 (Extremely Unlikely) to 7 (Extremely Likely). The participant is then asked how risky that behavior appears ranging from 1 (Not at all Risky) to 7 (Extremely Risky) and what the benefits are of that behavior from 1 (No Benefits at All) to 7 (Great Benefits). This self-report measure assesses the likelihood that a person will engage in five domains of risk behaviors (i.e., ethical, financial, health and safety, recreational, and social), as well as how risky the person perceives these behaviors to be and what benefits the person perceives will come from these behaviors. The scale is further broken into three subscales including: risk taking, risk perception, and risk benefits. Scores from the risk perception and risk benefits subscales combined to create a risk attitude score.
Change in impulsivity from baseline to 6 weeks | week 1 of study duration; week 6 of study duration
  The UPPS-P Impulsive Behavioral Scale assesses personality characteristics that lead to various impulsive like behaviors (e.g., Sensation Seeking's relationship with Extraversion). This measure consists of 59 items based on a 4-point Likert scales, ranging from 1 (Agree Strongly) to 4 (Disagree Strongly). This measure assesses impulsivity based on dimensions of the Five Factor Model of Personality and includes five sub-scales (i.e., Negative Urgency, Positive Urgency, [lack of] Premeditation, Sensation Seeking, and [lack of] Perseverance).

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Benning, PhD, Principal Investigator — University of Nevada, Las Vegas
Locations (1):
- University of Nevada Las Vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Undecided
If individual participant data is disseminated, it will include only data that has been de-identified. Specifically, only information regarding the effectiveness of the intervention will likely be reported. This could include statistics on urge-related behavior engagement, urge intensity, mental health symptoms, and personality factors.